CLINICAL TRIAL: NCT04161885
Title: A Randomized, Open Label Phase 3 Study Evaluating Safety and Efficacy of Venetoclax in Combination With Azacitidine After Allogeneic Stem Cell Transplantation in Subjects With Acute Myeloid Leukemia (AML) (VIALE-T)
Brief Title: A Study Evaluating Safety and Efficacy of Venetoclax in Combination With Azacitidine Versus Standard of Care After Allogeneic Stem Cell Transplantation (SCT) in Participants With Acute Myeloid Leukemia (AML)
Acronym: VIALE-T
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M19-063; 2023-507222-17-00 (Other: EU CT)
Record Dates: First submitted 2019-11-11; First posted 2019-11-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia (AML); Cancer
Keywords: Acute Myeloid Leukemia (AML); Venetoclax; Azacitidine; Stem Cell Transplantation (SCT); Best Support Care (BSC); Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1: Venetoclax + Azacitidine (AZA) + Best Supportive Care (Experimental): Participants will be administered various doses and dose regiments of venetoclax and AZA. Venetoclax will be administered once daily (QD) (Days 1-28) for up to 24 cycles, AZA QD on Days 1-5 of each 28-day cycle for up to 6 cycles and best supportive care (BSC) for 24 cycles (each cycle = 28 days)
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Other: Best Supportive Care (BSC)
- Part 2: Arm A - Venetoclax + Azacitidine (AZA) + BSC (Experimental): Participants will be administered with venetoclax and AZA at a dose level determined in Part 1 in addition to best supportive care (when required). Venetoclax will be administered once daily (QD) (Days 1-28) for up to 24 cycles, AZA QD on Days 1-5 of each 28-day cycle for up to 6 cycles and best supportive care (BSC) for 24 cycles (each cycle = 28 days).
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Other: Best Supportive Care (BSC)
- Part 2: Arm B - Best Supportive Care (BSC) (Experimental): Participants will receive treatment as prescribed by their physician according to the BSC for up to 24 cycles (1 cycle = 28 days)
  Interventions: Other: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Venetoclax — Tablet; Oral
  Other Names: ABT-199; GDC-0199; VENCLEXTA
  Arms: Part 1: Venetoclax + Azacitidine (AZA) + Best Supportive Care; Part 2: Arm A - Venetoclax + Azacitidine (AZA) + BSC
Drug: Azacitidine — Subcutaneous (SC) or intravenous (IV) injection
  Arms: Part 1: Venetoclax + Azacitidine (AZA) + Best Supportive Care; Part 2: Arm A - Venetoclax + Azacitidine (AZA) + BSC
Other: Best Supportive Care (BSC) — BSC is the best supportive care, without AML directed therapy, determined per the investigator and institutional guidelines.

SUMMARY:
The main objective of this study is to evaluate the efficacy of venetoclax in combination with azacitidine to improve Overall Survival (OS) in Acute Myeloid Leukemia (AML) participants compared to Best Supportive Care (BSC) when given as maintenance therapy following allogeneic stem cell transplantation (SCT).

This study will have 2 parts: Part 1 (Dose Confirmation), which may include participants who are greater than or equal to 18 years old; Part 2 (Randomization) which may include participants who are greater than or equal to 12 years old. During Part 1, recommended Phase 3 dose of venetoclax in combination with azacitidine will be determined and during Part 2, the efficacy and safety of venetoclax with azacitidine (Part 2 Arm A) will be compared with BSC (Part 2 Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old for Part 1 and, at least 12 years old for Part 2.
* Participant must be diagnosed with Acute Myeloid Leukemia (AML) by World Health Organization (WHO) criteria (2017) and either be planning for allogeneic stem cell transplantation or have received allogeneic stem cell transplantation within the past 60 days.
* Blast percentage in bone marrow before transplant must be < 10%.
* Blast count in peripheral blood must be "0" and Blast percentage in bone marrow must be < 5% after transplant.
* Participant meet adequate renal, hepatic and hematologic criteria as described in the protocol.
* Participants >= 17 years old must have a Karnofsky Performance Scale (KPS) score > 50 and participants between 12 to 16 years old must have a Lansky Play Performance Scale score > 40.

Exclusion Criteria:

* History of disease progression during prior treatment with venetoclax.
* History of any other malignancy within 2 years prior to study entry, except for: Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast; basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; previous malignancy confined and surgically resected (or treated with other modalities) with curative intent; Myelodysplastic Syndrome, Myeloproliferative neoplasm (only allowed if it transformed to AML and AML should be the indication for marrow transplantation).
* Participant has known infection with HIV or history of being positive for hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Presence of clinical or laboratory symptoms/signs of extramedullary myeloid malignancy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-Limiting Toxicities (DLTs) Following Administration of Venetoclax and Azacitidine (Part 1) | Up to the first treatment cycle (28 days)
  DLTs are any of the hematologic, nonhematologic toxicities, adverse events (AEs) occurring following administration of venetoclax and AZA as described in the protocol and evaluated by the Investigator and the sponsor.
Overall Survival (OS) (Part 2) | Up to 45 months after the first participant is randomized
  OS is defined as the number of days from the date of randomization to the date of death from any cause.

SECONDARY OUTCOMES:
Morphologic Relapse-Free Survival (RFS) (Part 2) | Up to 39 months after the first participant is randomized
  Morphologic relapse from AML defined as bone marrow blasts of >= 5% or reappearance of blasts in the peripheral blood not attributable to any other cause (e.g., bone marrow regeneration) in at least 2 peripheral blood samples at least one week apart or development of extramedullary disease after achieving a complete remission (CR) or complete remission with incomplete count recovery (CRi); or the date of death from any cause, whichever comes first as determined by Independent Review Committee (IRC).
Composite Relapse-Free Survival (RFS) (Part 2) | Up to 39 months after the first participant is randomized
  Morphologic relapse from AML, non-morphologic relapse from AML, which is defined as increase in disease burden determined by standard methods with reappearance or acquisition of new findings with or without change in anti-leukemic treatment per investigator decision due to cytogenetic abnormalities or change in molecular marker or measurable residual disease by multiparameter flow with sensitivity to at least 10^-3; or the date of death from any cause, whichever comes first as determined by IRC.
Graft-versus-Host Disease (GvHD)-free, Relapse Free Survival (GRFS) (Part 2) | Up to 39 months after the first participant is randomized
  GRFS is defined as number of days from the date of randomization to occurrence of disease relapse OR incidence of GvHD OR death from any cause.
Graft-versus-Host Disease (GvHD) Rate (Part 2) | Up to 39 months after the first participant is randomized
  GvHD rate is defined as grade 2 or higher for acute graft-versus-host disease (aGvHD) and moderate/severe for chronic graft-versus-host disease (cGvHD) assessed by investigator.
Change from Baseline in Physical Functioning as Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) (Part 2) | Up to 39 months after the first participant is randomized
  The EORTC-QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participantts rate items on a 4-point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Change From Randomization in Fatigue in Adult Participants (Part 2) | Up to 39 months after the first participant is randomized
  Fatigue is measured as Patient Reported Outcome (PRO) using Patient Reported Outcomes Measurement Information System (PROMIS) Cancer Fatigue SF 7a.
Measurable Residual Disease (MRD) Response Rate in Participants With MRD >= 10^-3 at Randomization (Part 2) | Up to 39 months after the first participant is randomized
  MRD conversion rate is defined as percentage of participants who convert to MRD < 10^-3 after initiation of treatment.
Time to Deterioration in Global Health Status (GHS)/Quality of Life (QoL) in Adult Participants (Part 2) | Up to 39 months after the first participant is randomized
  Time to deterioration defined as number of days from randomization to either deterioration of >= 5 points based on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) version 3 or death due to any cause.
Change in Patient Reported Signs, Symptoms and Impact of Acute Myeloid Leukemia (AML) as Measured by the European Quality-of-Life-5 Dimensional-5-Level (EQ-5D-5L) | Up to 39 months after the first participant is randomized
  The EQ-5D-5L is a generic preference instrument that has been validated in numerous population and has 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. These dimensions are measured on a 5-point scale: with higher scores representing better functioning/quality of life and greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (165):
- United States (43):
  - Arizona Oncology - Scottsdale - Cancer Transplant Institute /ID# 239711, Scottsdale, Arizona
  - University of Arizona Cancer Center - Tucson /ID# 242507, Tucson, Arizona
  - University of Arkansas for Medical Sciences /ID# 239804, Little Rock, Arkansas
  - City of Hope /ID# 213681, Duarte, California
  - UCHSC Anschultz Cancer Pavilion /ID# 215618, Aurora, Colorado
  - Colorado Blood Cancer Institute /ID# 215980, Denver, Colorado
  - Mayo Clinic /ID# 239710, Jacksonville, Florida
  - AdventHealth Medical Group Blood & Marrow Transplant at Orlando /ID# 213985, Orlando, Florida
  - Ann & Robert H Lurie Children's Hospital of Chicago /ID# 215840, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 215616, Chicago, Illinois
  - Loyola University Medical Ctr /ID# 215617, Maywood, Illinois
  - Indiana Blood & Marrow Transpl /ID# 215842, Indianapolis, Indiana
  - Duplicate_Ochsner Clinic Foundation-New Orleans /ID# 213834, New Orleans, Louisiana
  - University of Maryland, Baltimore /ID# 213855, Baltimore, Maryland
  - Massachusetts General Hospital /ID# 215765, Boston, Massachusetts
  - Karmanos Cancer Institute - Dresner Clinic /ID# 214581, Detroit, Michigan
  - Masonic Cancer Center /ID# 239492, Minneapolis, Minnesota
  - Mayo Clinic - Rochester /ID# 214685, Rochester, Minnesota
  - University of Mississippi Medical Center /ID# 239343, Jackson, Mississippi
  - The John Theurer Cancer /ID# 215251, Hackensack, New Jersey
  - Roswell Park Cancer Institute /ID# 217857, Buffalo, New York
  - Columbia University Medical Center /ID# 240875, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 240680, New York, New York
  - Weill Cornell Medical College /ID# 214887, New York, New York
  - Montefiore Medical Center - Moses Campus /ID# 241669, The Bronx, New York
  - University of North Carolina /ID# 215814, Chapel Hill, North Carolina
  - Wake Forest Univ HS /ID# 239210, Winston-Salem, North Carolina
  - UC Health - Cincinnati /ID# 239263, Cincinnati, Ohio
  - University Hospitals - Seidman Cancer Center /ID# 239260, Cleveland, Ohio
  - University of Oklahoma, Stephenson Cancer Center /ID# 215611, Oklahoma City, Oklahoma
  - Oregon Health and Science University /ID# 215874, Portland, Oregon
  - Penn State Hershey Medical Ctr /ID# 217120, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia - Main /ID# 215410, Philadelphia, Pennsylvania
  - Perelman Center for Advanced Medicine /ID# 214518, Philadelphia, Pennsylvania
  - Duplicate_Allegheny General Hospital /ID# 216756, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Ctr /ID# 213715, Pittsburgh, Pennsylvania
  - TriStar Centennial Medical Center /ID# 218750, Nashville, Tennessee
  - Texas Oncology - Medical City Dallas /ID# 216720, Dallas, Texas
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center /ID# 213735, Dallas, Texas
  - Texas Transplant Institute /ID# 214691, San Antonio, Texas
  - Virginia Commonwealth University Medical Center Main Hospital /ID# 239203, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center /ID# 214436, Seattle, Washington
  - Univ of Wisconsin Hosp/Clinics /ID# 216096, Madison, Wisconsin
- Australia (4):
  - The Kinghorn Cancer Centre /ID# 214660, Darlinghurst, New South Wales
  - Royal Adelaide Hospital /ID# 215678, Adelaide, South Australia
  - Peter MacCallum Cancer Ctr /ID# 214653, Melbourne, Victoria
  - The Alfred Hospital /ID# 240931, Melbourne, Victoria
- Brazil (4):
  - Hospital de Clinicas de Porto Alegre /ID# 215042, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho - Fundacao Doutor Amaral Carvalho /ID# 215145, Jaú, São Paulo
  - Hospital Nove de Julho /ID# 242359, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 239516, São Paulo
- Canada (5):
  - Vancouver Coastal Health Research Institute (VCHRI) /ID# 215363, Vancouver, British Columbia
  - University Health Network_Princess Margaret Cancer Centre /ID# 215344, Toronto, Ontario
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 214591, Montreal, Quebec
  - Royal Victoria Hospital / McGill University Health Centre /ID# 215253, Montreal, Quebec
  - Saskatoon Cancer Centre /ID# 238821, Saskatoon, Saskatchewan
- China (20):
  - Peking University People's Hospital /ID# 215551, Beijing, Beijing Municipality
  - Chinese PLA General Hospital /ID# 216287, Beijing, Beijing Municipality
  - Aerospace Center Hospital /ID# 217018, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital /ID# 215555, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital /ID# 218666, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University /ID# 216333, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 215553, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital /ID# 239401, Shenzhen, Guangdong
  - Henan Cancer Hospital /ID# 215554, Zhengzhou, Henan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Techno /ID# 215552, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 238373, Wuhan, Hubei
  - Xiangya Hospital Central South University /ID# 219025, Changsha, Hunan
  - Zhongda Hospital Southeast University /ID# 218926, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University /ID# 216605, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College /ID# 239098, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 239168, Nanchang, Jiangxi
  - Shanghai Changhai Hospital /ID# 216334, Shanghai, Shanghai Municipality
  - Tangdu Hospital of The Fourth Military Medical University, PLA /ID# 216282, Xi’an, Shanxi
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 215546, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 215550, Hangzhou, Zhejiang
- Czechia (4):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 214811, Brno, Brno-mesto
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 214814, Hradec Králové, Hradec Kralove
  - Fakultni Nemocnice Ostrava /ID# 239922, Ostrava, Ostrava-mesto
  - Ustav hematologie a krevni transfuze /ID# 215133, Prague
- France (8):
  - Duplicate_CHU de Nice - Hôpital Archet 1 /ID# 214056, Nice, Alpes-Maritimes
  - CHU de Besancon - Jean Minjoz /ID# 241171, Besançon, Doubs
  - Duplicate_CHU Bordeaux - Hopital Haut Leveque /ID# 214055, Pessac, Gironde
  - CHRU Lille - Hopital Claude Huriez /ID# 217916, Lille, Nord
  - CHU de Nantes, Hotel Dieu -HME /ID# 214060, Nantes, Pays de la Loire Region
  - Hôpital Saint-Louis /ID# 214054, Paris
  - AP-HP - Hopital Saint-Antoine /ID# 216957, Paris
  - Hopital Pitie Salpetriere /ID# 241072, Paris, Île-de-France Region
- Germany (8):
  - Universitaetsklinik Heidelberg /ID# 216623, Heidelberg, Baden-Wurttemberg
  - Klinikum Augsburg /ID# 239583, Augsburg, Bavaria
  - Universitaetsklinikum Wuerzburg /ID# 215212, Würzburg, Bavaria
  - Universitaetsklinikum Muenster /ID# 215213, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 214244, Dresden, Saxony
  - Universitaetsklinikum Leipzig /ID# 245892, Leipzig, Saxony
  - Universitaetsklinikum Halle (Saale) /ID# 239585, Halle
  - Medizinische Hochschule Hannover /ID# 214243, Hanover
- Greece (3):
  - General Hospital of Athens Evangelismos /ID# 238810, Athens, Attica
  - University General Hospital Attikon /ID# 238812, Athens, Attica
  - University General Hospital of Patras /ID# 238811, RION Patras Achaia
- Debreceni Egyetem-Klinikai Kozpont /ID# 241123, Debrecen, Hajdú-Bihar, Hungary
- Israel (7):
  - Schneider Children's Medical Center /ID# 224326, Petah Tikva, Central District
  - Rambam Health Care Campus /ID# 214507, Haifa, H_efa
  - Hadassah Medical Center-Hebrew University /ID# 218697, Jerusalem, Jerusalem
  - Sheba Medical Center /ID# 239571, Ramat Gan, Tel Aviv
  - The Chaim Sheba Medical Center /ID# 214305, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 214508, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 214509, Petah Tikva
- Italy (6):
  - IRCCS Ospedale San Raffaele /ID# 214311, Milan, Milano
  - Istituto Europeo Di Oncologia /ID# 242579, Milan, Milano
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 216148, Turin, Piedmont
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 254964, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 214910, Rome, Roma
  - ASST degli Spedali Civili di Brescia /ID# 215997, Brescia
- Japan (26):
  - Anjou Kousei Hospital /ID# 215857, Anjo-shi, Aichi-ken
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital /ID# 215679, Nagoya, Aichi-ken
  - University of Fukui Hospital /ID# 253383, Yoshida-gun, Fukui
  - Kyushu University Hospital /ID# 215285, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 252293, Fukushima, Fukushima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital /ID# 217522, Hiroshima, Hiroshima
  - Hokkaido University Hospital /ID# 215937, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital /ID# 215388, Kobe, Hyōgo
  - Hyogo Medical University Hospital /ID# 215389, Nishinomiya-shi, Hyōgo
  - Kanazawa University Hospital /ID# 242955, Kanazawa, Ishikawa-ken
  - Imamura General Hospital /ID# 215688, Kagoshima, Kagoshima-ken
  - Tokai University Hospital /ID# 250086, Isehara, Kanagawa
  - Kanagawa Cancer Center /ID# 215029, Yokohama, Kanagawa
  - Kyoto University Hospital /ID# 243209, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 214670, Sendai, Miyagi
  - Okayama University Hospital /ID# 214842, Okayama, Okayama-ken
  - Osaka Metropolitan University Hospital /ID# 215227, Osaka, Osaka
  - Kindai University Hospital /ID# 214917, Osakasayama-shi, Osaka
  - Jichi Medical University Saitama Medical Center /ID# 216092, Saitama-shi, Saitama
  - Jichi Medical University Hospital /ID# 216091, Shimotsuke-shi, Tochigi
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital /ID# 215939, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital /ID# 242639, Chuo-ku, Tokyo
  - Toranomon Hospital /ID# 215311, Minato-ku, Tokyo
  - National Center for Child Health and Development /ID# 242479, Setagaya-ku, Tokyo
  - Keio University Hospital /ID# 243549, Shinjuku-ku, Tokyo
  - Yamagata University Hospital /ID# 253304, Yamagata, Yamagata
- South Korea (4):
  - Seoul National University Hospital /ID# 214891, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 214893, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 239087, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 214892, Seoul, Seoul Teugbyeolsi
- Spain (7):
  - Hospital Clinic de Barcelona /ID# 215108, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 240397, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 215107, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 218102, Madrid
  - Hospital Universitario La Paz /ID# 218103, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 215463, Seville
  - Hospital Clinico Universitario de Valencia /ID# 215106, Valencia
- Switzerland (2):
  - Duplicate_Universitätsspital Basel /ID# 215892, Basel, Canton of Basel-City
  - University Hospital Zurich /ID# 215891, Zurich, Canton of Zurich
- Taiwan (6):
  - National Taiwan University Hospital /ID# 215245, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 215197, Kaohsiung City
  - China Medical University Hospital /ID# 215198, Taichung
  - Taichung Veterans General Hospital /ID# 239288, Taichung
  - Taipei Veterans General Hosp /ID# 239289, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 215319, Taoyuan
- United Kingdom (7):
  - Hammersmith Hospital /ID# 215665, London, England
  - Gartnavel General Hospital /ID# 215663, Glasgow, Glasgow City
  - University College London Hospital /ID# 215662, London, Greater London
  - University Hospitals Birmingham NHS Foundation Trust /ID# 215120, Birmingham
  - King's College Hospital NHS Foundation Trust /ID# 215338, London
  - The Royal Marsden NHS Foundation Trust /ID# 215124, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 248359, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M19-063